CLINICAL TRIAL: NCT02341703
Title: Letrozole-metformin Versus Letrozole-metformin-pioglitazone in PCO Clomiphene Citrate Resistant Women
Brief Title: Ovulation Induction in Clomiphene Citrate Resistant PCO Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Abdel Fattah, assistant professor of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University Hospital
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Polycystic Ovary Syndrome; Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- letrozole-metformin group (Active Comparator): this group will receive letrozole 2.5 mg daily from day 3 of the cycle and for 5 days + metformin 500 mg three times daily from the first day of the cycle and continuous for three months unless pregnancy occurred. treatment will continue for 3 cycles unless pregnancy occurred.
  for this group: transvaginal ultrasound will monitor follicular enlargement laboratory investigations in the form of day 3 FSH, LH, TSH and serum testosterone will be done day 12 E2 day 21 serum progesterone
  Interventions: Drug: letrozole-metformin; Radiation: transvaginal ultrasound; Other: laboratory investigations
- letrozole-metformin-pioglitazone group (Active Comparator): this group will receive letrozole 2.5 mg daily from day 3 of the cycle and for 5 days + (metformin 850 mg + pioglitazone 15 mg) once daily from the first day of the cycle and for 10 days. treatment will continue for 3 cycles unless pregnancy occurred.
  for this group: transvaginal ultrasound will monitor follicular enlargement laboratory investigations in the form of day 3 FSH, LH, TSH and serum testosterone will be done day 12 E2 day 21 serum progesterone
  Interventions: Drug: letrozole-metformin-pioglitazone; Radiation: transvaginal ultrasound; Other: laboratory investigations

INTERVENTIONS:
Drug: letrozole-metformin — letrozole 2.5 mg will be given daily from day 3 of the cycle for 5 days + metformin 500 mg three times daily continuously for 3 months unless pregnancy occurred
  Other Names: femara-cidophage
  Arms: letrozole-metformin group
Drug: letrozole-metformin-pioglitazone — letrozole will be given daily from day 3 of the cycle for 5 days + (metformin 850 mg + pioglitazone 15 mg) from the first day of the cycle for 10 days.
  Other Names: femara- bioglita plus
  Arms: letrozole-metformin-pioglitazone group
Radiation: transvaginal ultrasound — transvaginal ultrasound will be done from day 10 of the cycle and every other day for monitoring of follicular enlargement.
Other: laboratory investigations — day 3: FSH, LH, TSH, and total testosterone day 12 serum E2 day 21 serum progesterone

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 5-10% of women in childbearing age. Hyperinsulinemia contributes to chronic anovulation commonly encountered in women with PCOS. The first choice therapy is clomiphene citrate (CC). In CC resistant cases, the American College of Obstetrics and Gynecology (ACOG) recommends the use of insulin sensitizer metformin. Other insulin sensitizing agents include rosiglitazone and pioglitazone. Pioglitazone is said to improve fertility and ovulation in patients with PCOS.CC may be associated with poor endometrial thickening due to its antiestrogenic effect. Letrozole may improve this condition. In this study we will compare the effect of combined letrozole-metformin with that of combined letrozole-pioglitazone in ovulation induction in CC-resistant PCOS women

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 5-10% of women in childbearing age. Hyperinsulinemia contributes to chronic anovulation commonly encountered in women with PCOS. The first choice therapy is clomiphene citrate (CC). In CC resistant cases, the ACOG recommends the use of insulin sensitizer metformin. Other insulin sensitizing agents include rosiglitazone and pioglitazone. Pioglitazone is said to improve fertility and ovulation in patients with PCOS. CC has a long half-life (2 weeks), and this may have a negative effect on the cervical mucus and endometrium, leading to discrepancy between ovulation and conception rates. There has been a search for a compound capable of inducing ovulation but devoid of the adverse antiestrogenic effects of CC. recent studies have suggested that letrozole, an aromatase inhibitor, does not possess the adverse antiestrogenic effects of CC and is associated with higher pregnancy rates than CC treatment in patients with PCOS.

In this study the investigators shall compare the effect of combined letrozole-metformin with that of combined letrozole-metformin-pioglitazone in ovulation induction in CC-resistant PCOS women.This will be a prospective comparative clinical trial in which 2 groups of women will be generated (groups A and B) using the sealed envelopes randomization method.Group A (50 women) will receive: letrozole 2.5 mg/day from 3rd day of the cycle for 5 days and (pioglitazone 15 mg + metformin 850 mg) once daily from 1st day of the cycle for 10 days. Group B (50 women) will receive letrozole 2.5 mg/day from 3rd day of the cycle for 5 days and metformin 500 mg three times daily from continuously untill pregncy occurrs. Ovulation will be monitored by vaginal ultrasound and serum estrogen and progesterone.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old
* PCOS infertile women resistant to CC for 3 cycles

Exclusion Criteria:

* Presence of medical disorders as diabetes, hypertension, cardiac problems, liver or kidney diseases, hyperprolactinemia or thyroid dysfunction
* Use of gonadotropins before
* Previous ovarian drilling
* Presence of urinary symptoms especially bloody urine

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
ovulation rate | 6 months

SECONDARY OUTCOMES:
pregnancy rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdel Fattah Abdel Moety, lecturer, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine, Cairo University, Cairo, Cairo Governorate, Egypt